CLINICAL TRIAL: NCT04037774
Title: Comparision of Different Doses of Dexmedetomidine With Low Dose Bupivacaine in Selective Spinal Anesthesia for Transurethral Resection of Prostate in Elderly Males.
Brief Title: Comparision of Different Doses of Dexmedetomidine With Low Dose Bupivacaine in Selective Spinal Anesthesia.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Services Institute of Medical Sciences, Pakistan (Other Government)
Responsible Party: Principal Investigator, dr. sana siddiq, professor of anesthesiology, Services Institute of Medical Sciences, Pakistan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: simsanesthesia
Record Dates: First submitted 2019-05-05; First posted 2019-07-30 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Drug Effect
Keywords: analgesia,; spinal block; dexmedetomidine; bupivacaine; selective spinal anesthesia
MeSH Terms: conditions — Agnosia | interventions — Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: randomized control design
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- dex 5microgram (Active Comparator): this group of patients is given total 2ml solution intrathecally, 1ml of 5mg local anesthetic i.e 0.5% hyperbaric bupivacaine and 1ml of 5micrograms of dexmedetomidine.
  Interventions: Drug: Dexmedetomidine
- dex 10microgram (Active Comparator): this group of patients is given total 2ml solution intrathecally, 1ml of 5mg local anesthetic i.e 0.5% hyperbaric bupivacaine and 1ml of 10micrograms of dexmedetomidine.
  Interventions: Drug: Dexmedetomidine
- placebo (Placebo Comparator): this group of patients is given total 2ml solution intrathecally, 1ml of 5mg local anesthetic i.e 0.5% hyperbaric bupivacaine and 1ml of placebo.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Dexmedetomidine — comparision of different doses of dexmedetomidine used intrathecally
  Arms: dex 10microgram; dex 5microgram
Other: placebo — addition of placebo with local anesthetic to create a control group
  Arms: placebo

SUMMARY:
The charactereistics of a spinal block varies with the dose of local anaesthetic and the adjuvant used. Literature review did not show comparison of different doses of dexmedetomidine with low-dose bupivacaine in saddle block. The rationale of this study is to determine an optimum dose of dexmedetomidine which in combination with low dose bupivacaine would provide satisfactory block with hemodynamic stability. This would be beneficial for patients scheduled for turp, as these pts are mostly elderly with various comorbidities.

DETAILED DESCRIPTION:
SYNOPSIS:

Comparison of different doses of intra-thecal dexmedetomidine as an additive to low-dose bupivacaine(5mg) in selective spinal anesthesia for transurethral resection of prostate in elderly patients.

Introduction:

Most patients scheduled for Transurethral Resection of the Prostate Gland are elderly and usually present with cardiovascular, endocrine, renal, cerebral or respiratory diseases thereby increasing their risk for surgery and anaesthesia. Spinal anesthesia is the technique of choice in transurethral resection of prostate . The major problem of spinal technique is risk of hypotension. In spinal anesthesia due to sympathetic blockade, there is vasodilatation leading to diminished venous return which is the main contributory factor for hypotension. 1 Selective spinal anesthesia , commonly known as saddle block, is defined as "the practice of employing minimal doses of intrathecal agents so that only the nerve roots supplying a specific area and only the modality that require to be anesthetized are affected." Thus, Selective spinal anesthesia is more appropriate in elderly patients3 Saddle block paralyzed pelvic muscles and sacral nerve roots. As lower level of block is achieved, hemodynamic derangement is less and fluid requirement is also less. So there is minimum chance of circulatory overload1 but may provide insufficient surgical anaesthesia.5and also may not achieve an extended duration of postoperative analgesia.2 Dexmedetomidine is a highly selective alpha2 adrenoceptor (α2-AR) agonist recently introduced to anaesthesia practice. It produces dose-dependent sedation, anxiolysis and analgesia (involving spinal and supraspinal sites) without respiratory depression7 intrathecal Dex has been used as an adjuvant to different local anesthetics in humans with various doses ranging from 2.5 to 15 micrograms [2,3,9-15] resulting in improving the quality of sensory and motor blockade and increasing their duration and decreasing the dose of local anesthetic used intrathecal Dex has been used as an adjuvant to different local anesthetics in humans with various doses ranging from 2.5 to 15 micrograms [2,3,9-15] resulting in improving the quality of sensory and motor blockade and increasing their duration and decreasing the dose of local anesthetic used intrathecal Dex has been used as an adjuvant to different local anesthetics in humans with various doses ranging from 2.5 to 15 micrograms, resulting in improving the quality of sensory and motor blockade and increasing their duration and decreasing the dose of local anesthetic used.4

RATIONALE:

The charactereistics of a spinal block varies with the dose of local anaesthetic and the adjuvant used. Literature review did not show comparison of different doses of dexmedetomidine with low-dose bupivacaine in saddle block. The rationale of this study is to determine an optimum dose of dexmedetomidine which in combination with low dose bupivacaine would provide satisfactory block with hemodynamic stability. This would be beneficial for patients scheduled for transurethral resection of prostate, as these patients are mostly elderly with various comorbidities.

Objective:

To evaluate and compare the effects of Two doses of intra-thecal dexmedetomidine (5 and 10 µgrams) with 5mg hyperbaric bupivacaine, and 5mg hyperbaric bupivacaine alone in saddle block for ,

* onset and regression of sensory block times,
* peak sensory block,
* hemodynamic changes,
* adequate surgical conditions
* duration of effective post-operative analgesia

Operational definations:

MEAN ARTERIAL PRESSURE:

The arithmetic mean of the blood pressure in the arterial part of the circulation, it is calculated by adding the systolic pressure reading to two times the diastolic reading and dividing the sum by 3.

record arterial blood pressure and mean heart rate for both groups.

Adequate surgical conditions:

Sensory block height till T12 and adequate relaxation of pelvic floor muscles will be considered optimal surgical conditions.

Post-operative analgesia:

Time from intrathecal drug administration till demand of first rescue analgesia is considered as effective post-opertaive analgesic period.

onset of sensory block: Time from intrathecal drug injection till achievement of highest sensory block level would be labelled as onset of sensory block.

Regression of sensory block:

Time from intrathecal drug injection till two segment sensory regression from peak sensory level .

Hypothesis: higher doses of dexmedetomdine with low dose bupivacaine provide more prolongation of effective post-operative analgesia, as compared too low doses.

Materials and Methods:

Study design: single blind prospective randomized control trial. Setting: After approval from ethical committee, this study will be conducted at the Department Of Anesthesiology and Surgical Intensive Care Unit , services Hospital Lahore.

Duration of study: The proposed study will be completed in six months after approval of synopsis from services institute of medical sciences.

Sample size:

Sample size is calculated by taking mean time to 2 segment regression in minutes from following data, 116±20.1 vs 130 ± 15.5 At significance level of alpha 5% , confidence level 90% power of study 80% estimated sample size is 25 for each group.

Inclusion criteria:

Male gender, age between 50 and 70 years old and Patients' physical status by the American Society of Anesthesiologist (ASA): ASA class I, II and III

Exclusion criteria:

Contraindications of spinal anesthesia, Patients who were taking α2-adrenergic agonist or antagonist therapy, Patients who were having labile hypertension, uncontrolled cardiac disease, heart block/dysrhythmia, autoimmune disorders, Communication difficulties, e.g. mental retardation or deafness and Allergy to the drug or local anesthetics.

Study procedures:

Seventy five elderly male patients in the age group between 55 and 75 years and American Society of Anesthesiologists Grade I-III undergoing Transuretheral resection of prostate will be included in this study. Using a computer-generated random number table, patients will be enrolled in one of the two groups, Group I: will receive 5 mg of 0.5% hyperbaric bupivacaine hydrochloride( 1ml) with 5 micro grams of dexmedetomidine (1ml). Total drug volume will be 2ml.

Group II : will receive 10 μg of dexmedetomidine hydrochloride(1ml) combined with 5mg of 0.5% hyperbaric bupivacaine hydrochloride. Total drug volume will be 2ml.

Group III: will receive 5mg of 0.5% hyperbaric bupivacaine(1ml) with 1ml of Normal sline as placebo.

Each patient will recieve an appropriate randomised number allocated to his group according to the number, sealed and packed inside opaque covers and labelled with the project title, investigators' name and the randomisation number..

Standard monitoring including electrocardiogram , pulse oximetry and noninvasive blood pressure will be attached to the patients upon their arrival to the operating room. Baseline parameters will be recorded, and monitoring will be initiated. Intravenous access will be secured using 18Gauge cannula. patients will be made to position is sitting position for institution of saddle block. Complete aseptic precautions including cleaning with povidone iodine and draping will be performed. The L3/L4 or L4/L5 intervertebral space will be located. The skin overlying the intervertebral space after identification will be anesthetized with 3 ml of 2% lidocaine using a size 22Gauge hypodermic needle. Lumbar puncture will be performed using a 23 or 25Gauge pencil point spinal needle to inject the study agent intrathecally. After testing the backflow of cerebrospinal fluid, the intrathecal injectate will be given over approximately ten seconds. The spinal needle will then withdrawn, and a light dressing will be placed over the puncture site.

Patients will remain in sitting position for atleast 10 minutes, then patients will be made to lie supine. The level of sensory block will be determined using the hub of a sterile 22-gauge needle in the midline, and dermatomal level will be assessed every 2 min from completion of injection until the assessed sensory level remained stable for four consecutive assessments. Testing will be conducted every 10 min thereafter until two-segment regression will be noticed. Further testing will be performed at 20 min intervals in the recovery room until regression of 2 segments from peak sensory levels . Systolic blood pressure, diastolic blood pressure and heart rate will be recorded every 3 min for the first 15 min following spinal anaesthesia, and then every 5 min until the end of surgery. Hypotension (Systolic blood-pressure <90 mmHg or 30% decrease from the baseline) and bradycardia (Heart rate <45 beats/min) will be treated with Intravenous bolus of phenylephrine 50 micrograms alliquots and atropine 0.6 milligram, respectively. Adverse effects such as nausea, vomiting, shivering, pruritus, respiratory depression, and transient neurological symptoms will be recorded. The duration of surgery will be noted. The patients would be instructed to tell the staff nurse whenever they felt the need for an analgesic. The staff nurse will note the time to first analgesic request from the patient within 24 hours after surgery. Toradol Intravenous 30 mg and paracetamol Intravenous 1gram would be the postoperative rescue analgesics.

Statistics: Statistical analysis will be done by SPSS 20. Demographic data will be expressed as mean±SD. Mean time to Onset of sensory block, two segment regression of sensory block and duration of analgesia between groups will be analysed by one way ANOVA. Haemodynamic measures will be analysed by repeated measures ANOVA. Intergroup comparison of Level of sensory block will be done by Mann Whitney U test. A p value <0.05 will be taken as significant.

ELIGIBILITY:
Inclusion Criteria:

Male gender Age between 50 and 70 years old Patients' physical status by the American Society of Anesthesiologist (ASA): ASA class I, II and III

Exclusion Criteria:

Contraindications of spinal anesthesia, Patients who were taking α2-adrenergic agonist or antagonist therapy, Patients who were having labile hypertension, uncontrolled cardiac disease, heart block/dysrhythmia, autoimmune disorders, Communication difficulties, e.g. mental retardation or deafness Allergy to the drug or local anesthetics.

Min Age: 20 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — only in transuretheral resection of prostate patients.
Enrollment: 75 (Estimated)
Dates: Start 2019-09-02 (Estimated); Primary Completion 2019-11-01 (Estimated); Study Completion 2019-11-01 (Estimated)

PRIMARY OUTCOMES:
duration of post-operative analgesia | upto 6months
  duration the patient remains pain free from administration of drug.

SECONDARY OUTCOMES:
peak sensory level | upto 6 months
  peak sensory level attained after drug administration
2 segment regression | upto 6 months
  time to achieve 2 segment regression from the time at which patient achieved peak sensory level
side effects | upto 6 months
  side effects noted during and after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Services Institute of Medical Sciences, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No